CLINICAL TRIAL: NCT04509687
Title: Feasibility Study of Training Endoscopists to Perform On-site Rapid Cytological Evaluation for Endoscopic Ultrasound-guided Fine-needle Aspiration of Solid Pancreatic Lesions
Brief Title: Training Endoscopists to Perform On-site Rapid Cytological Evaluation for EUS-FNA of Solid Pancreatic Lesions
Acronym: EUS-FNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, chief of the gastroenterology, Changhai Hospital
Other Study IDs: ROSE
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — pancreatic sample acquired from EUS-FNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In China, there is a serious shortage of pathologists who can perform on-site cytological diagnosis. As a result, there are few centers that can conduct ROSE in China, which limits the diagnostic accuracy of EUS-FNA to a certain extent. Previous research reports on whether endoscopists could be trained for ROSE were controversial, which may be related to the lack of standardization of the training of endoscopists. There is no training program for training endoscopists to systematically process pathological specimens, operate microscopes, read the adequacy of cytological specimens, and evaluate the atypia of cytological specimens in China. Therefore, our center intends to carry out a training for endoscopists to compare the improvement of endoscopists' ROSE operating ability before and after the training, and to evaluate the practice of each endoscopist to perform on-site rapid cytology specimens of solid pancreatic lesions.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years
2. diagnosis or suspected of solid pancreatic mass based on previous imaging examination;
3. EUS-FNA is achievable.
4. signed informed consent letter

Exclusion Criteria:

1. pregnant female
2. pancreatic cystic lesions
3. anticoagulant/antiplatelet therapy cannot be suspended
4. unable or refuse to provide informed consent
5. coagulopathy (platelet count <50 ×103/uL, international normalized ration >1.5）
6. severe cardiopulmonary dysfunction that cannot tolerate intravenous anesthesia
7. with history of mental disease
8. other medical conditions that are not suitable for EUS-FNA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to involve 60 patients with solid pancreatic lesion, with trained endoscopists performing ROSE in the procedure of EUS-FNA
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of endoscopists for interpretation of cytologic specimen adequacy and primary diagnosis of malignancy | 10 months
  The interpretation results of endoscopists will be compared with that of cytopathologist.

SECONDARY OUTCOMES:
The results of standard specimens-processing, microscope-operating training on endoscopists | 3 months
  Comparison of the score that endoscopists are graded before and after the standard training

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China